CLINICAL TRIAL: NCT00698074
Title: Diastolic Ventricular Interaction and the Effects of Biventricular Pacing in Hypertrophic Cardiomyopathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 05/Q2709/64
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 1 (Experimental): Cardiac Resynchronisation Therapy
  Interventions: Device: Cardiac Resynchronisation Therapy

INTERVENTIONS:
Device: Cardiac Resynchronisation Therapy — Biventricular Pacemaker Implant

SUMMARY:
The primary aim of this study will be to assess whether Biventricular pacing improves exercise capacity, and Quality of Life in patients with symptomatic drug resistant Non-Obstructive Hypertrophic Cardiomyopathy, using a Biventricular pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Hypertrophic Cardiomyopathy,

Exclusion Criteria:

* Rhythm other than normal sinus Left ventricular outflow tract gradient greater than 30mmHg Inability to exercise v02 max greater than 70% of predicted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Department Cardiovascular Medicine, University of Birmingham, Birmingham, West Midlands, United Kingdom